CLINICAL TRIAL: NCT06923683
Title: The Effectiveness of a Treatment for Social Cognition Disorders (T-ScEmo) in Patients With Acquired Brain Injury and Comorbid Neuropsychiatric Problems
Brief Title: Treatment for Social Cognition Disorders (T-ScEmo) in Patients With Acquired Brain Injury and Comorbid Neuropsychiatric Problems
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ggz Oost Brabant (Other)
Collaborators: Maastricht University (Other); UMC Groningen, Groningen, the Netherlands (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-ScEmo SCED
Record Dates: First submitted 2025-02-28; First posted 2025-04-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-01

CONDITIONS: Acquired Brain Injury; Neuropsychiatric Symptoms
MeSH Terms: conditions — Brain Injuries | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- There is only one arm in this study, since it is a SCED. (Experimental)
  Interventions: Behavioral: Treatment for social cognition disorders (T-ScEmo)

INTERVENTIONS:
Behavioral: Treatment for social cognition disorders (T-ScEmo) — T-ScEmo is an evidence-based, multifaceted treatment protocol for poor social cognition and emotion regulation impairments in patients with ABI. T-ScEmo is implemented as standard practice in the Netherlands. In total, the treatment consists of 20 1-hour sessions. The treatment is divided into extended psychoeducation for patient and proxy and 3 modules, including emotion perception (module 1), perspective taking and understanding social information (module 2), and goal-directed social behavior (module 3). These three modules are interdependent and strengthen each other. Therefore, the developers strongly recommend to offer all three modules. The presence of a proxy is required in the first psycho-education session and during the third module. The first and second modules are invariant (10 sessions together), but in the third module, therapists can adjust the content to individual needs and personal goals.

SUMMARY:
Acquired brain injury (ABI) can lead to a wide range of physical, cognitive, emotional, and social problems. In the recent years, more research has been conducted to examine the impact of ABI on social cognition. Approximately 13%-40% of patients with ABI experience difficulties with social cognition. Social cognition refers to the cognitive processes involved in perceiving, interpreting, and responding to social information. When these processes are disrupted, patients may struggle to (1) understand social situations, (2) interpret the emotions and intentions of others, and (3) respond appropriately in social interactions. This not only results in reduced social engagement for ABI patients, but also places a burden on relationships and proxies. Therefore, it is important to effectively treat social cognition problems in ABI patients.

To date, only a few treatment studies aimed at improving social cognition have been conducted. In 2017, a multifaceted treatment for impairments in social cognition and emotion regulation (T-ScEmo) is developed, which was proven effective in improving multiple aspects of social cognition and emotion regulation. T-ScEmo is now considered as an evidence-based treatment for patients with traumatic brain injury and social cognition problems. However, ABI patients and comorbid neuropsychiatric problems have been excluded in most studies exploring the treatment of social cognition problems after ABI. It is important that the effect of T-ScEmo in this particular group is examined, since 25%-88% of the ABI patients experience neuropsychiatric problems. Comorbidities are thus very prevalent in this ABI population.

Unfortunately, up till now there are no studies examining the effect of T-ScEmo in patients with ABI, comorbid neuropsychiatric problems and social cognition problems. Therefore, the aim of the present study is threefold:

1. To examine the effect of a treatment for impairments in social cognition and emotion regulation (T-ScEmo) on social cognition problems;
2. To examine the effect of T-ScEmo on social interaction, communication and neuropsychiatric behavioral problems;
3. To examine the effect of T-ScEmo on quality of partner relationship in patients with ABI and comorbid psychiatric problems.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* have an established and documented history of ABI and current neuropsychiatric problems. When patients are referred to our institution, a team of clinical neuropsychologists, psychiatrists, and a high-educated nurse estimate whether patients meet these criteria by using a transdiagnostic tool.
* have social cognition problems. These impairments in social cognition are established by defective scores on the Facial Expression of Emotion-Stimuli and Tests (FEEST) and/or (if available) frontal lesions visible on computed tomographic scan/magnetic resonance image, indicating higher risk on social behavioral problems. The FEEST is already used in standard care.
* are at least 6 months post-injury to avoid the effects of spontaneous recovery.
* are between 18 and 70 years.
* have a significant other/proxy to fill in questionnaires and participate in the treatment. A life partner (persons living together in an intimate relationship, either married or unmarried) is preferred. When patients don't have a life partner, they are asked to bring an adult proxy (a close friend or family member) with whom they have frequent contact in daily life, preferably someone who already knew the patient from before the ABI.

Exclusion Criteria:

* not being able to receive the T-ScEmo treatment, for example due to severe cognitive impairment
* not speaking the Dutch language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Social functioning - Social Functioning Scale (SFS) | From enrollment to follow-up, approximately 12 months.
  Functioning in social situations is measured by using a Social Functioning Scale (SFS), where patients and proxies rate the patient's functioning in social situations on a 10-point scale from 1 ("not at all") to 10 ("entirely"). The following question will be asked to patients and proxies: "How satisfied are you today with your (or your partner's) functioning in social situations?" Higher scores indicate more satisfaction.
Neuropsychiatric behavior problems - Neuropsychiatric behavior Problems Scale (NPS) | From enrollment to follow-up, approximately 12 months.
  Neuropsychiatric behavior problems are measured by using a Neuropsychiatric behavior Problems Scale (NPS), where patients and proxies rate the patient's neuropsychiatric behavior problems on a 10-point scale from 1 ("not at all") to 10 ("entirely"). The following question will be asked to patients and proxies: "To what extent did you (or your partner) experience neuropsychiatric behavioral problems today?". 'Neuropsychiatric behavioral problems' refer to the neuropsychiatric problems that the client is (most) affected by (e.g. irritability, aggression, disinhibition, depression, anxiety).
  Higher scores indicate more neuropsychiatric problems.
Relationship quality - Relationship Quality Scale (RQS) | From enrollment to follow-up, approximately 12 months.
  Relationship quality is measured by using the Relationship Quality Scale (RQS), where patients and proxies rate the quality of their relationship on a 10-point scale from 1 ("not at all") to 10 ("entirely"). Higher scores indicate more satisfaction.

SECONDARY OUTCOMES:
Executive functioning (social scales) | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Dysexecutive Questionnaire - Social scales (DEX-Soc-self; DEX-Soc-proxy) will be filled out by participant and proxy. The DEX subscales 'Meta cognition' (items 2, 5, 12, 16, 20), 'Social convention' (items 9, 12, 13, 20), and 'Behavioral emotional self-regulation' (items 3, 7, 8) will be filled out. The items are scored on a 4-point scale (0 = never to 4 = very often), with higher scores indicating more problems.
Social monitoring | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Brock's Adaptive Functioning Questionnaire Social monitoring scale (BAFQ-SMself, BAFQ-SM-proxy) will be filled out by participant and proxy. The items are scored on a 5-point scale (1 = almost never to 5 = almost ever), with higher scores indicating more problems.
Empathy | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The IRI (Interpersonal Reactivity Index) will be filled out by the participant. The IRI is a 28-item multidimensional scale that measures empathy. The scale measures both the cognitive and affective aspects of empathy. The IRI consists of 4 subscales, each containing 7 items. Higher scores indicate a higher level of empathy.
  The Brock's Adaptive Functioning Questionnaire Empathy scale (BAFQ-Emp-self, BAFQ-Emp-proxy) will be filled out by participant and proxy. The items are scored on a 5-point scale (1 = almost never to 5 = almost ever), with higher scores indicating more problems.
Neuropsychiatric problems | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Neuropsychiatrische Vragenlijst-Questionnaire (NPI-Q) will be filled out by the proxy. The NPI-Q is a validated questionnaire, aimed at inventorying neuropsychiatric symptoms that have occurred in the past month. For each domain, the answer is initially given as "Yes" (present) or "No" (absent). If the answer is "No," the informant proceeds to the next question. If the answer is "Yes," the informant assesses both the severity of the symptoms that occurred in the past month (three-point scale) and the psychological burden it caused for him or her (six-point scale). The NPI-Q provides a severity rating and an assessment of the emotional burden for each reported symptom, as well as summed total scores for Severity and Emotional Burden. Higher scores indicate more problems.
Cognitive Communication | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The the La Trobe Questionnaire (LCQ-S / LCQ-O) will be filled out by participant and proxy. The LCQ-S is a 30-item self-report questionnaire that assesses perceived communication quality in patients with ABI. Items of the LCQ-O are the same as those that appear in de LCQ-S, except they are phrased in the third person. Higher scores indicate more problems.
Marital Satisfaction | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Dutch Marital Satisfaction and Communication Questionnaire (DMSCQ) will be filled out by participant and proxy. The DMSCQ is a 16-item questionnaire that disentangles marital satisfaction, negative communication and open communication on a 7-point scale ("not at all applicable" to "highly applicable")
Caregiver strain | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Caregiver Strain Index (CSI) will be filled out by the proxy to detect caregiver strain. The CSI is a 13-item questionnaire with dichotomous yes/no answers. Higher scores indicate more problems.
Recognition of facial affect | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The FEEST (Sixty faces test) will be administered to test the recognition of facial affect. Participants are presented with 60 photographs of faces displaying the various primary emotions (happiness, sadness, fear, angst, disgust, and surprise), with 10 faces of each primary emotion. The photographs are shown for 3 seconds. Higher scores indicate a better performance.
Mental state attribution | At baseline, post-treatment (22-29 weeks), and follow-up (approximately 1 year after baseline)
  The Cartoon test will be administered to test mental state attribution. The Cartoon test incorporates 12 cartoons displaying humorous situations. Higher scores indicate a better performance.

OTHER OUTCOMES:
Other neuropsychological tests | At baseline
  Other neuropsychological tests are used to assess possible effects of cognitive (dis)functioning on effectiveness of the treatment, neuropsychological tests on attention, executive functioning, and memory will be administered before treatment: Trail Making Test (TMT) A + B, TMT B/A; BADS Zoo-map; 15-word test.

CONTACTS AND LOCATIONS:
Locations (1):
- GGZ Oost Brabant, Boekel, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No